CLINICAL TRIAL: NCT01301456
Title: A Phase 1, Double-blind, Placebo-controlled, Randomized, Parallel Group Study To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Pf-04856883 In Adult Female Subjects With Type 2 Diabetes Mellitus
Brief Title: Single-Dose And Multiple-Dose Safety And Tolerability Study Of PF-04856883 In Type 2 Diabetic Adult Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1111002
Record Dates: First submitted 2011-02-09; First posted 2011-02-23 (Estimated); Results first posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases
Keywords: Phase 1; Type 2 Diabetes; CVX-096
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (13):
- Treatment Arm 1 (Stage 1A) (Placebo Comparator)
  Interventions: Biological: Placebo
- Treatment Arm 2 (Stage 1A) (Experimental)
  Interventions: Biological: PF-04856883
- Treatment Arm 3 (Stage 1A) (Experimental)
  Interventions: Biological: PF-04856883
- Treatment Arm 4 (Stage 1A) (Experimental)
  Interventions: Biological: PF-04856883
- Treatment Arm 5 (Stage 1B) (Placebo Comparator)
  Interventions: Biological: Placebo
- Treatment Arm 6 (Stage 1B) (Experimental)
  Interventions: Biological: PF-04856883
- Treatment Arm 7 (Stage 1B) (Experimental)
  Interventions: Biological: PF-04856883
- Treatment Arm 8 (Stage 1B) (Experimental)
  Interventions: Biological: PF-04856883
- Treatment Arm 9 (Stage 2) (Placebo Comparator)
  Interventions: Biological: Placebo
- Treatment Arm 10 (Stage 2) (Experimental)
  Interventions: Biological: PF-04856883
- Treatment Arm 11 (Stage 2) (Experimental)
  Interventions: Biological: PF-04856883
- Treatment Arm 12 (Stage 2) (Experimental)
  Interventions: Biological: PF-04856883
- Treatment Arm 13 (Stage 2) (Experimental)
  Interventions: Biological: PF-04856883

INTERVENTIONS:
Biological: Placebo — Single subcutaneous injection of placebo
  Arms: Treatment Arm 1 (Stage 1A)
Biological: PF-04856883 — Single subcutaneous injection of PF-04856883
  Other Names: CVX-096
  Arms: Treatment Arm 2 (Stage 1A)
Biological: PF-04856883 — Single subcutaneous injection of PF-04856883
  Other Names: CVX-096
  Arms: Treatment Arm 3 (Stage 1A)
Biological: PF-04856883 — Single subcutaneous injection of PF-04856883
  Other Names: CVX-096
  Arms: Treatment Arm 4 (Stage 1A)
Biological: Placebo — Single subcutaneous injection of placebo
  Arms: Treatment Arm 5 (Stage 1B)
Biological: PF-04856883 — Single subcutaneous injection of PF-04856883
  Other Names: CVX-096
  Arms: Treatment Arm 6 (Stage 1B)
Biological: PF-04856883 — Single subcutaneous injection of PF-04856883
  Other Names: CVX-096
  Arms: Treatment Arm 7 (Stage 1B)
Biological: PF-04856883 — Single subcutaneous injection of PF-04856883
  Other Names: CVX-096
  Arms: Treatment Arm 8 (Stage 1B)
Biological: Placebo — Multiple weekly subcutaneous injections of placebo for 3 weeks
  Other Names: CVX-096
  Arms: Treatment Arm 9 (Stage 2)
Biological: PF-04856883 — Multiple weekly subcutaneous injections of PF-04856883 for 3 weeks
  Other Names: CVX-096
  Arms: Treatment Arm 10 (Stage 2)
Biological: PF-04856883 — Multiple weekly subcutaneous injections of PF-04856883 for 3 weeks
  Other Names: CVX-096
  Arms: Treatment Arm 11 (Stage 2)
Biological: PF-04856883 — Multiple weekly subcutaneous injections of PF-04856883 for 3 weeks
  Other Names: CVX-096
  Arms: Treatment Arm 12 (Stage 2)
Biological: PF-04856883 — Multiple weekly subcutaneous injections of PF-04856883 for 3 weeks
  Other Names: CVX-096
  Arms: Treatment Arm 13 (Stage 2)

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of PF-04856883 (CVX-096) in adult female subjects with Type 2 diabetes mellitus on high dose of metformin.

ELIGIBILITY:
Inclusion Criteria:

* History of Type 2 diabetes and currently being treated with high dose metformin
* BMI between 22.0 and 40.0 kg/m2
* HbA1c between 7.0-10.0%
* Fasting C-peptide >1.21 ng/mL

Exclusion Criteria:

* History of clinically significant chronic conditions other than Type 2 diabetes not well controlled by either diet or medications
* Treatment with anti-diabetic therapies other than metformin
* History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody
* Males or women of childbearing potential

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 84 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Profil Institute for Clinical Research, Inc., Chula Vista, California
  - Elite Research Institute, Miami, Florida
  - Comprehensive Phase One (A Division of Comprehensive NeuroScience, Inc.), Miramar, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - ICON Clinical Pharmacology, LLC, Omaha, Nebraska
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - Healthcare Discoveries LLC d/b/a ICON Development Solutions, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1111002&StudyName=Single-Dose%20And%20Multiple-Dose%20Safety%20And%20Tolerability%20Study%20Of%20PF-04856883%20In%20Type%202%20Diabetic%20Adult%20Females%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data for reporting arm Placebo 1a and 1b in stage 1 was planned to be pooled during analysis, as per protocol. Study consisted of two stages: stage 1 and stage 2. Participants were enrolled and randomized for stage 1 and stage 2 separately.
Groups:
- Stage 1: PF-04856883 Placebo: Participants received placebo matched to PF-04856883 subcutaneously injection once on Day 1 in Stage 1.
- Stage 1: PF-04856883 4 mg: Participants received PF-04856883 4 milligram (mg) subcutaneous injection once on Day 1 in Stage 1.
- Stage 1: PF-04856883 8 mg: Participants received PF-04856883 8 mg subcutaneous injection once on Day 1 in Stage 1.
- Stage 1: PF-04856883 12 mg: Participants received PF-04856883 12 mg subcutaneous injection once on Day 1 in Stage 1.
- Stage 1: PF-04856883 18 mg: Participants received PF-04856883 18 mg subcutaneous injection once on Day 1 in Stage 1.
- Stage 1: PF-04856883 24 mg: Participants received PF-04856883 24 mg subcutaneous injection once on Day 1 in Stage 1.
- Stage 1: PF-04856883 36 mg: Participants received PF-04856883 36 mg subcutaneous injection once on Day 1 in Stage 1.
- Stage 2: Placebo: Participants received placebo matched to PF-04856883 subcutaneous injection on Day 1, 8, 15 and 22 respectively in Stage 2.
- Stage 2: PF-04856883 12 mg: Participants received single dose of PF-04856883 12 mg subcutaneous injection on Day 1, 8, 15 and 22 respectively in Stage 2.
- Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg: Participants received single dose of PF-04856883 12 mg, 12 mg, 24 mg, 24 mg subcutaneous injection on Day 1, 8, 15 and 22 respectively in Stage 2.
- Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg: Participants received single dose of PF-04856883 8 mg, 8 mg, 16 mg, 24 mg subcutaneous injection on Day 1, 8, 15 and 22 respectively in Stage 2.
- Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg: Participants received single dose of PF-04856883 12 mg, 20 mg, 28 mg, 36 mg subcutaneous injection on Day 1, 8, 15 and 22 respectively in Stage 2.
Period: Stage 1
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Started | 15 | 5 | 6 | 6 | 7 | 5 | 8 | 0 | 0 | 0 | 0 | 0
Received Treatment | 15 | 5 | 6 | 6 | 7 | 5 | 7 | 0 | 0 | 0 | 0 | 0
Completed | 15 | 5 | 5 | 6 | 6 | 5 | 7 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5 | 7 | 7 | 6
Received Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5 | 7 | 7 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5 | 7 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized.
Groups:
- Stage 1: PF-04856883 4 mg: Participants received PF-04856883 4 mg subcutaneous injection once on Day 1 in Stage 1.
- Total: Total of all reporting groups
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg | Total
Number analyzed (Participants) | 15 | 5 | 6 | 6 | 7 | 5 | 8 | 7 | 5 | 7 | 7 | 6 | 84
Age, Customized [Number; unit: participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 64 years | 15 | 3 | 5 | 4 | 6 | 4 | 6 | 6 | 5 | 4 | 7 | 6 | 71
  >=65 years | 0 | 2 | 1 | 2 | 1 | 1 | 2 | 1 | 0 | 3 | 0 | 0 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 5 | 6 | 6 | 7 | 5 | 8 | 7 | 5 | 7 | 7 | 6 | 84
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose (Day 50) that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Stage 1: Baseline up to Day 29; Stage 2: Baseline up to Day 50
Population: The safety population included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 15 | 5 | 6 | 6 | 7 | 5 | 7 | 7 | 5 | 7 | 7 | 6
participants
  SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AE | 8 | 1 | 0 | 2 | 4 | 3 | 4 | 4 | 5 | 5 | 5 | 5

2. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Description: Physical examination included examination of general appearance, head, ears, eyes (including fundoscopy), nose, mouth, throat, neck (including thyroid), skin, breast (optional), cardiac, respiratory, gastrointestinal, musculoskeletal and neurological systems.
Time Frame: Stage 1: Baseline up to Day 29; Stage 2: Baseline up to Day 50
Population: The safety population included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Groups:
- Stage 1: PF-04856883 36mg Single Dose: Participants received subcutaneous injection of PF-04856883 4 mg by a 4-week follow up period in Stage 1
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36mg Single Dose | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 15 | 5 | 6 | 6 | 7 | 5 | 7 | 7 | 5 | 7 | 7 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiograms (ECG)
Description: ECG parameters included pulse rate (PR) interval, QRS interval, corrected QT interval using Bazett's formula (QTcB) and corrected QT interval using Fridericia's formula (QTcF). ECG criteria of clinically significant concern were 1) PR interval: greater than equal to (>=) 25 percent (%) increase when baseline greater than (>)200 milliseconds (msec); or increase >=50% when baseline less than or equal to (<=200) msec; 2) QRS interval: >=25% increase when baseline >100 msec; >=50% increase when baseline <= 100 msec; 3) QTCF interval: QTc interval using Fridericia's formula (QTcF interval) and Bazett's formula (QTcB interval): absolute value 450 - <480 msec, 480 - <500 msec >=500; absolute change 30 - <60, >=60 msec. The number of participants with potentially clinically significant ECG findings at any visit were reported. IFB = increase from baseline.
Time Frame: Stage 1: Baseline up to Day 29; Stage 2: Baseline up to Day 50
Population: The safety population included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 15 | 5 | 6 | 6 | 7 | 5 | 7 | 7 | 5 | 7 | 7 | 6
participants
  Maximum PR Interval IFB: >=25 or 50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Maximum QTcB Interval IFB: 30-<60 msec | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
  Maximum QTcF Interval IFB: 30-<60 msec | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Criteria for vital signs abnormalities: sitting/supine systolic pulse rate less than (<) 40 beats per minute (bpm) or greater than (>) 120 bpm, standing/supine systolic pulse < 40 bpm or > 140 bpm, systolic blood pressure of >=30 millimeters of mercury (mmHg) change from baseline and systolic blood pressure <90 mmHg, diastolic blood pressure >=20 mmHg change from baseline and diastolic blood pressure <50 mm Hg.
Time Frame: Stage 1: Baseline up to Day 29; Stage 2 : Baseline up to Day 50
Population: The safety population included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 15 | 5 | 6 | 6 | 7 | 5 | 7 | 7 | 5 | 7 | 7 | 6
participants | 15 | 5 | 6 | 6 | 7 | 5 | 7 | 7 | 5 | 7 | 7 | 6

5. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Measurements
Description: Following parameters were analyzed for laboratory examination: Hematology: hemoglobin, hematocrit, red blood cell (RBC) <0.8*lower limit of the reference range (LLRR); leukocytes <0.6*LLRR or >1.5*ULRR; platelet count <0.5*LLRR or >1.75*upper limit of the reference range (ULRR); total neutrophils (absolute [abs]), lymphocytes (abs) <0.8*LLRR or >1.2*ULRR; eosinophils (abs), basophils (abs), monocytes (abs) >1.2*ULRR; chemistry (total bilirubin, direct bilirubin, indirect bilirubin >1.5*ULRR; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase >3*ULRR, albumin, total protein <0.8*LLRR or >1.2*ULRR; blood urea nitrogen (BUN), creatinine >1.3*ULRR; glucose (fasting) <0.6*LLRR or >1.5*ULRR; uric acid >1.2* ULRR; sodium <0.95*LLRR or >1.05*ULRR; potassium, chloride, bicarbonate, calcium <0.9*LLRR or >1.1*ULRR. Urinalysis: Urine white blood cell (WBC), Urine RBC =>20/ high-power field (HPF).
Time Frame: Stage 1: Baseline up to Day 29; Stage 2: Baseline up to Day 50
Population: The safety population included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 15 | 5 | 6 | 6 | 7 | 5 | 7 | 7 | 5 | 7 | 7 | 6
participants | 15 | 5 | 6 | 6 | 7 | 4 | 6 | 7 | 5 | 7 | 7 | 6

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-04856883: Stage 1
Time Frame: predose (0 hour), 1, 6, 12, 24, 48, 72, 120, 168, 336, 504, 672 hours postdose on Day 1
Population: Pharmacokinetic (PK) parameter analysis population included all randomized participants who had received at least one dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg
Number analyzed (Participants) | 5 | 6 | 6 | 7 | 5 | 7
nanogram per milliliter (ng/mL) | 181.2 (85) | 324.7 (61) | 793.7 (65) | 1855 (66) | 1776 (21) | 2006 (52)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-04856883: Stage 2
Time Frame: predose (0 hour), 1, 6, 12, 24, 48, 72, 120, 168, 336 hours postdose on Day 1; predose (0 hour), 1, 2, 6, 24, 48, 72, 120, 168, 336, 504, 672 hours postdose on Day 22
Population: PK parameter analysis population included all randomized participants who had received at least one dose of study treatment and had at least 1 of the PK parameters of interest. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 5 | 7 | 7 | 6
ng/mL
  Day 1 (n =5, 7, 7, 6) | 1369 (17) | 1203 (20) | 1027 (29) | 1407 (29)
  Day 22 (n =5, 7, 5, 6) | 1802 (33) | 2757 (26) | 3030 (42) | 3046 (24)

8. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04856883: Stage 1
Time Frame: predose (0 hour), 1, 6, 12, 24, 48, 72, 120, 168, 336, 504, 672 hours postdose on Day 1
Population: PK parameter analysis population included all randomized participants who had received at least one dose of study treatment and had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: hour
Arm/Group | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg
Number analyzed (Participants) | 5 | 6 | 6 | 7 | 5 | 7
hour | 168 [72.0 to 336] | 120 [48.0 to 168] | 120 [48.0 to 168] | 120 [48.0 to 120] | 120 [72.0 to 168] | 122 [120 to 168]

9. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04856883: Stage 2
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 5 | 7 | 7 | 6
hour
  Day 1 (n =5, 7, 7, 6) | 336 [336 to 336] | 336 [335 to 336] | 335 [24.1 to 336] | 336 [336 to 336]
  Day 22 (n =5, 7, 5, 6) | 48.0 [24.0 to 72.0] | 72.0 [0.000 to 72.0] | 72.0 [48.0 to 72.1] | 60.0 [0.000 to 120]

10. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC [0 - ∞]) of PF-04856883: Stage 1
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: predose (0 hour), 1, 6, 12, 24, 48, 72, 120, 168, 336, 504, 672 hours postdose on Day 1
Population: PK parameter analysis population included all randomized participants who had received at least one dose of study treatment and had at least 1 of the PK parameters of interest. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg
Number analyzed (Participants) | 3 | 3 | 4 | 5 | 3 | 3
nanogram*hour per milliliter (ng*hr/mL) | 44920 (112) | 95190 (76) | 295200 (46) | 527100 (53) | 711300 (13) | 652000 (50)

11. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Time Tau (AUCtau) of PF-04856883: Stage 2
Description: Area under the serum concentration-time curve from time 0 to tau (AUCtau), where tau was the dosing interval of 168 hours.
Time Frame: predose (0 hour), 1, 6, 12, 24, 48, 72, 120, 168 hours postdose Day 1; predose (0 hour), 1, 2, 6, 24, 48, 72, 120, 168 hours postdose Day 22
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 5 | 7 | 7 | 6
ng*hr/mL
  Day 1 (n =5, 7, 7, 6) | 85370 (38) | 99780 (41) | 89390 (35) | 91130 (27)
  Day 22 (n =5, 7, 5, 6) | 269000 (32) | 377400 (28) | 396300 (28) | 430500 (23)

12. Secondary Outcome: Apparent Clearance (CL/F) of PF-04856883: Stage 1
Description: It was calculated by dividing dose with AUC (0 - ∞) where AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). Outcome measure was planned to be analyzed in Stage 1 only.
Time Frame: predose (0 hour), 1, 6, 12, 24, 48, 72, 120, 168, 336, 504, 672 hours postdose on Day 1
Population: PK parameter analysis population included all randomized participants who had received at least one dose of study treatment and had at least 1 of the PK parameters of interest. Here, 'N' signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per hour (mL/hr)
Arm/Group | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg
Number analyzed (Participants) | 3 | 3 | 4 | 5 | 3 | 3
milliliter per hour (mL/hr) | 89.14 (84) | 84.08 (59) | 40.60 (68) | 34.13 (35) | 33.73 (14) | 55.32 (42)

13. Secondary Outcome: Apparent Clearance (CL/F) of PF-04856883: Stage 2
Description: It was calculated by dividing dose with AUC (0 - ∞) where AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). Outcome measure was planned to be analyzed in Stage 2 only. Data was not estimable if values were below the limit of quantification.
Time Frame: predose (0 hour), 1, 2, 6, 24, 48, 72, 120, 168, 336, 504, 672 hours postdose on Day 22
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 5 | 7 | 7 | 6
mL/hr | 44.67 (28) | NA (NA) — Data was not estimable since values were below the limit of quantification. | NA (NA) — Data was not estimable since values were below the limit of quantification. | NA (NA) — Data was not estimable since values were below the limit of quantification.

14. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-04856883: Stage 1
Time Frame: predose (0 hour), 1, 6, 12, 24, 48, 72, 120, 168, 336, 504, 672 hours postdose on Day 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter (mL)
Arm/Group | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg
Number analyzed (Participants) | 3 | 3 | 4 | 5 | 3 | 3
milliliter (mL) | 18760 (90) | 21710 (59) | 9191 (51) | 7127 (40) | 8437 (17) | 10010 (67)

15. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-04856883: Stage 2
Time Frame: predose (0 hour), 1, 2, 6, 24, 48, 72, 120, 168, 336, 504, 672 hours postdose on Day 22
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 5 | 7 | 7 | 6
mL | 9550 (29) | NA (NA) — Data was not estimable since values were below the limit of quantification. | NA (NA) — Data was not estimable since values were below the limit of quantification. | NA (NA) — Data was not estimable since values were below the limit of quantification.

16. Secondary Outcome: Terminal Elimination Half- Life (t1/2) of PF-04856883: Stage 1
Time Frame: predose (0 hour), 1, 6, 12, 24, 48, 72, 120, 168, 336, 504, 672 hours postdose on Day 1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 3 | 3
hour | 146.3 (13.614) | 179.7 (14.572) | 147.0 (18.520) | 133.8 (23.936) | 173.7 (7.0238) | 131.6 (45.883)

17. Secondary Outcome: Terminal Elimination Half-life (t1/2) of PF-04856883: Stage 2
Time Frame: predose (0 hour), 1, 2, 6, 24, 48, 72, 120, 168, 336, 504, 672 hours postdose on Day 22
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 5 | 5 | 4 | 5
hour | 149.4 (21.870) | 135.0 (43.980) | 143.8 (20.565) | 145.0 (37.000)

18. Secondary Outcome: Change From Baseline in Post-prandial Glucose Area Under the Curve (AUC) After Mixed Meal Tolerance Test (MMTT) at Day 3 and 8: Stage 1
Description: Change from baseline in post-prandial area under the plasma glucose concentration time curve as determined by standardized MMTT. Linear trapezoidal method was used to compute AUC
Time Frame: Baseline, Day 3 and 8
Population: Pharmacodynamic analysis population included all enrolled participants who had received at least 1 dose of study treatment and have at least 1 pharmacodynamic parameter. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: milligram*hour per deciliter (mg*hr/dL)
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg
Number analyzed (Participants) | 15 | 5 | 6 | 6 | 7 | 5 | 7
milligram*hour per deciliter (mg*hr/dL)
  Baseline (n =15, 5, 6, 6, 7, 5, 7) | 656.35 (114.496) | 834.03 (158.952) | 712.11 (88.942) | 796.14 (208.733) | 660.64 (110.833) | 652.20 (48.707) | 636.57 (119.662)
  Change at Day 3 (n =15, 5, 5, 6, 7, 5, 6) | 7.72 (89.366) | 77.82 (125.011) | -89.38 (58.909) | -101.47 (31.725) | -68.05 (111.431) | -141.27 (15.975) | -153.04 (41.501)
  Change at Day 8 (n =15, 5, 5, 6, 7, 5, 6) | -4.82 (75.396) | 10.37 (158.368) | 0.85 (125.384) | -82.51 (48.898) | -28.36 (61.456) | -123.43 (68.219) | -39.60 (85.256)

19. Secondary Outcome: Change From Baseline in Post-prandial Glucose Area Under the Curve (AUC) After Mixed Meal Tolerance Test (MMTT) at Day 3, 15, 24, 29 and 50: Stage 2
Description: as for outcome 18
Time Frame: Baseline, Day 3, 15, 24, 29 and 50
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 7 | 5 | 7 | 7 | 6
mg*hr/dL
  Baseline (n =7, 4, 7, 7, 6) | 606.49 (158.249) | 811.36 (131.145) | 756.17 (240.430) | 800.66 (206.776) | 723.57 (220.872)
  Change at Day 3 (n =7, 4, 5, 6, 5) | 44.41 (74.405) | -97.03 (55.692) | -103.00 (118.759) | -98.38 (114.644) | -68.52 (153.127)
  Change at Day 15 (n =7, 4, 6, 6, 6) | -18.48 (50.874) | -265.64 (89.889) | -293.04 (163.074) | -254.54 (144.897) | -240.65 (252.349)
  Change at Day 24 (n =7, 4, 7, 6, 5) | -6.20 (46.238) | -146.61 (78.863) | -207.12 (89.687) | -242.35 (231.302) | -121.13 (258.528)
  Change at Day 29 (n =7, 4, 7, 6, 5) | 30.08 (59.490) | -55.43 (74.973) | -157.54 (88.652) | -192.97 (185.056) | -106.58 (171.297)
  Change at Day 50 (n =7, 3, 6, 6, 6) | 50.26 (81.717) | -48.82 (80.733) | -33.77 (250.859) | -125.06 (217.403) | -23.99 (123.611)

20. Secondary Outcome: Change From Baseline in Insulin Area Under the Curve (AUC) After Mixed Meal Tolerance Test (MMTT) at Day 3 and 8: Stage 1
Description: Change from baseline in post-prandial plasma insulin AUC under the plasma insulin concentration versus time curve as determined by standardized MMTT. Linear trapezoidal method was used to compute AUC.
Time Frame: Baseline, Day 3 and 8
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: milliUnit*hour per liter (mU*hr/L)
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg
Number analyzed (Participants) | 15 | 5 | 6 | 6 | 7 | 5 | 7
milliUnit*hour per liter (mU*hr/L)
  Baseline (n =15, 5, 6, 6, 7, 5, 7) | 222.18 (139.981) | 227.07 (142.547) | 210.80 (95.536) | 235.84 (130.071) | 105.34 (19.118) | 257.73 (127.358) | 283.59 (156.831)
  Change at Day 3 (n =15, 5, 5, 6, 7, 5, 6) | 68.79 (115.555) | 22.99 (32.706) | 35.09 (57.093) | 12.15 (54.495) | 59.06 (94.643) | 83.82 (70.182) | 13.72 (98.682)
  Change at Day 8 (n =15, 4, 5, 6, 7, 5, 6) | 34.23 (103.279) | 22.05 (89.419) | 39.96 (38.941) | -50.51 (40.624) | 38.04 (15.736) | -0.36 (50.674) | 1.08 (47.135)

21. Secondary Outcome: Change From Baseline in Insulin Area Under the Curve (AUC) After Mixed Meal Tolerance Test (MMTT) at Day 3, 15, 24, 29 and 50: Stage 2
Description: as for outcome 20
Time Frame: Baseline, Day 3, 15, 24, 29 and 50
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mU*hr/L
Arm/Group | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 7 | 5 | 7 | 7 | 6
mU*hr/L
  Baseline (n =7, 5, 7, 7, 6) | 175.26 (62.218) | 176.65 (76.040) | 267.29 (111.497) | 162.96 (111.688) | 190.64 (83.945)
  Change at Day 3 (n =7, 5, 7, 7, 6) | 38.32 (62.135) | 13.29 (55.764) | 19.50 (134.651) | 27.99 (32.655) | 87.67 (124.052)
  Change at Day 15 (n =7, 5, 7, 6, 6) | -16.77 (20.530) | -39.16 (42.930) | -10.07 (172.044) | -51.69 (77.925) | -24.36 (85.633)
  Change at Day 24 (n =7, 4, 7, 6, 6) | 0.23 (55.174) | -15.19 (38.900) | 6.87 (184.830) | 4.18 (51.903) | 60.11 (189.287)
  Change at Day 29 (n =7, 5, 7, 6, 5) | 8.25 (55.799) | 3.98 (11.218) | 12.71 (115.095) | -1.61 (85.866) | 15.70 (38.476)
  Change at Day 50 (n =7, 5, 7, 6, 5) | 8.14 (29.909) | -16.64 (33.133) | -57.14 (116.193) | 49.27 (81.874) | -26.78 (81.518)

22. Secondary Outcome: Change From Baseline in C-Peptide Area Under the Curve (AUC) After Mixed Meal Tolerance Test (MMTT) at Day 3 and 8: Stage 1
Description: Change from baseline in post-prandial area under the plasma C-peptide concentration time curve as determined by standardized MMTT. Linear trapezoidal method was used to compute AUC.
Time Frame: Baseline, Day 3 and 8
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg
Number analyzed (Participants) | 15 | 5 | 6 | 6 | 7 | 5 | 7
ng*hr/mL
  Baseline (n =15, 5, 6, 6, 7,5, 7) | 15.53 (5.332) | 16.63 (7.743) | 16.43 (4.306) | 16.80 (5.711) | 10.64 (1.156) | 16.17 (4.531) | 18.37 (7.395)
  Change at Day 3 (n =15, 5, 5, 6, 7, 5, 6) | 2.15 (3.653) | 0.69 (1.465) | 1.65 (4.958) | 1.05 (1.885) | 4.30 (4.102) | 5.34 (2.584) | 2.34 (4.333)
  Change at Day 8 (n =15, 4, 5, 6, 7, 5, 6) | 0.79 (2.864) | 1.06 (1.806) | 0.83 (1.651) | -2.74 (1.380) | 1.70 (1.544) | -0.45 (2.883) | -0.38 (1.565)

23. Secondary Outcome: Change From Baseline in C-Peptide Area Under the Curve (AUC) After Mixed Meal Tolerance Test (MMTT) at Day 3, 15, 24, 29 and 50: Stage 2
Description: as for outcome 22
Time Frame: Baseline, Day 3, 15, 24, 29 and 50
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 7 | 5 | 7 | 7 | 6
ng*hr/mL
  Baseline (n =7, 5, 7, 7, 6) | 13.47 (4.315) | 14.59 (4.205) | 15.63 (4.293) | 11.74 (5.210) | 14.14 (5.211)
  Change at Day 3 (n =7, 5, 7, 7, 6) | 1.68 (2.182) | 1.89 (4.705) | 0.50 (4.757) | 3.16 (1.613) | 3.49 (4.452)
  Change at Day 15 (n =7, 5, 7, 6, 6) | -1.65 (1.493) | -1.55 (2.821) | -1.92 (6.930) | -0.17 (4.135) | -0.50 (4.871)
  Change at Day 24 (n =7, 4, 7, 6, 6) | 0.55 (3.518) | 0.71 (4.312) | -0.99 (6.220) | 1.63 (2.994) | 1.21 (5.784)
  Change at Day 29 (n =7, 5, 7, 6, 5) | 0.10 (3.864) | -0.07 (2.545) | -0.59 (4.144) | 0.59 (2.733) | 0.41 (2.090)
  Change at Day 50 (n =7, 5, 7, 6, 5) | -0.17 (1.978) | -1.83 (2.015) | -4.10 (5.265) | 1.06 (1.474) | -2.90 (3.711)

24. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Day 2, 4, 6, 15, 22 and 29: Stage 1
Time Frame: Baseline, Day 2, 4, 6, 15, 22 and 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Groups:
- Stage 2: PF-04856883 36 mg: Participants received PF-04856883 36 mg subcutaneous injection once on Day 1 in Stage 1.
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 2: PF-04856883 36 mg
Number analyzed (Participants) | 15 | 5 | 6 | 6 | 7 | 5 | 7
milligram per deciliter (mg/dL)
  Baseline (n =15, 5, 6, 6, 7, 5, 7) | 161.67 (27.102) | 219.60 (44.557) | 171.17 (23.752) | 174.00 (48.949) | 168.57 (38.336) | 145.60 (21.606) | 158.14 (35.362)
  Change at Day 2 (n =15, 5, 6, 6, 7, 5, 7) | 3.13 (11.807) | 13.60 (32.393) | -18.67 (21.011) | -20.50 (20.433) | -22.14 (34.090) | -35.00 (12.369) | -29.71 (30.804)
  Change at Day 4 (n =15, 5, 5, 6, 7, 5, 6) | 2.73 (17.161) | 19.60 (35.683) | -12.40 (17.358) | -10.33 (15.744) | -30.71 (13.841) | -27.00 (8.803) | -28.33 (21.942)
  Change at Day 6 (n =15, 5, 4, 6, 7, 5, 7) | 18.80 (29.547) | 26.40 (32.377) | 10.25 (29.056) | -8.33 (27.156) | -6.29 (15.850) | -16.80 (19.176) | -16.14 (22.319)
  Change at Day 15 (n =15, 5, 5, 6, 6, 5, 7) | 12.13 (32.822) | -13.80 (46.949) | 23.80 (56.857) | 19.33 (16.476) | 8.00 (21.223) | 3.40 (27.309) | -2.71 (16.530)
  Change at Day 22 (n =14, 4, 5, 6, 6, 5, 7) | 11.00 (28.205) | 23.75 (61.163) | 33.40 (76.064) | 11.17 (26.446) | 2.17 (15.065) | 1.20 (18.847) | -0.57 (13.377)
  Change at Day 29 (n =14, 5, 5, 6, 7, 5, 7) | 22.00 (33.439) | 1.60 (27.763) | 27.80 (29.575) | 0.33 (16.978) | 1.57 (21.220) | -3.80 (22.643) | -2.29 (19.551)

25. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Day 2, 4, 6, 8, 22, 23, 25, 27, 30, 36 and 43: Stage 2
Time Frame: Baseline, Day 2, 4, 6, 8, 22, 23, 25, 27, 30, 36 and 43
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 7 | 5 | 7 | 7 | 6
mg/dL
  Baseline (n =7, 5, 7, 7, 6) | 148.00 (33.317) | 186.80 (23.059) | 191.14 (56.153) | 187.29 (45.756) | 158.50 (18.447)
  Change at Day 2 (n =5, 4, 7, 7, 5) | 3.00 (15.281) | -26.75 (15.108) | -15.14 (21.217) | -23.43 (35.142) | -10.40 (18.461)
  Change at Day 4 (n =5, 5, 7, 6, 6) | 7.60 (6.427) | -14.80 (24.284) | -14.86 (48.657) | -20.33 (22.818) | -1.50 (27.384)
  Change at Day 6 (n =7, 4, 7, 7, 6) | -1.71 (40.240) | 5.75 (14.080) | -44.86 (38.451) | -8.00 (42.942) | -15.83 (8.909)
  Change at Day 8 (n =6, 5, 7, 5, 6) | 2.50 (17.627) | 4.20 (19.967) | -37.43 (42.383) | 2.60 (73.449) | 24.50 (47.618)
  Change at Day 22 (n =7, 4, 7, 6, 6) | 13.29 (15.294) | -4.25 (13.817) | -39.57 (25.468) | -14.17 (38.270) | -0.33 (51.181)
  Change at Day 23 (n =7, 4, 6, 6, 5) | 7.71 (23.894) | -27.25 (27.293) | -40.33 (18.327) | -17.50 (73.519) | -24.00 (29.967)
  Change at Day 25 (n =7, 5, 6, 6, 5) | 13.43 (13.113) | -16.60 (43.443) | -44.67 (27.667) | -23.33 (52.936) | -16.20 (36.513)
  Change at Day 27 (n =7, 5, 6, 6, 5) | 8.57 (21.110) | -21.60 (15.821) | -37.33 (17.963) | -34.67 (35.803) | 12.00 (71.039)
  Change at Day 30 (n =7, 5, 7, 6, 5) | 2.43 (12.739) | -14.20 (17.908) | -22.29 (26.171) | -9.33 (32.898) | 15.40 (37.964)
  Change at Day 36 (n =6, 5, 7, 6, 6) | -10.50 (32.415) | 0.40 (37.846) | 1.86 (25.373) | -5.83 (32.009) | 27.67 (59.594)
  Change at Day 43 (n =7, 5, 5, 6, 6) | 18.71 (22.552) | 12.80 (29.064) | 13.20 (17.254) | -1.17 (41.787) | 8.33 (18.991)

26. Secondary Outcome: Change From Baseline in 24 Hours Glucose Normalized Area Under the Curve (NAUC) Profile at Day 30: Stage 2
Description: A normalized area under the curve (NAUC) were computed by dividing the AUC by the amount of time between the last time point captured and the first time point captured.
Time Frame: Baseline, Day 30
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 7 | 5 | 7 | 7 | 6
mg/dL
  Baseline (n =7, 5, 7, 7 ,6) | 166.19 (35.437) | 212.43 (52.764) | 205.56 (51.907) | 202.43 (38.900) | 186.13 (33.839)
  Change at Day 30 (n =7, 5, 7, 6 ,5) | 172.36 (38.825) | 191.20 (43.953) | 172.24 (48.067) | 174.08 (41.437) | 192.87 (58.037)
Statistical Analysis 1: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg; Day 30; Test type: Superiority or Other; p = 0.219, Mixed meal tolerance test; Least square (LS) mean = -21.16, 80% CI 2-sided [-43.26 to 0.93], Standard Error of Mean 16.766
Statistical Analysis 2: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg; Day 30; Test type: Superiority or Other; p = 0.034, Mixed meal tolerance test; LS mean = -34.18, 80% CI 2-sided [-54.20 to -14.16], Standard Error of Mean 15.189
Statistical Analysis 3: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg; Day 30; Test type: Superiority or Other; p = 0.044, Mixed meal tolerance test; LS mean = -33.67, 80% CI 2-sided [-54.50 to -12.84], Standard Error of Mean 15.806
Statistical Analysis 4: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg; Day 30; Test type: Superiority or Other; p = 0.857, Mixed meal tolerance test; LS mean = -2.93, 80% CI 2-sided [-24.16 to 18.31], Standard Error of Mean 16.111

27. Secondary Outcome: Percent Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Day 29 and 50: Stage 2
Description: HbA1c is a measure of the glycosylated hemoglobin. Change (measured as percent): HbA1c at observation minus HbA1c at baseline. Outcome measure was planned to analyzed only for Stage 2.
Time Frame: Baseline, Day 29 and 50
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 7 | 5 | 7 | 7 | 6
percent
  Day 29 (n =7, 5, 7, 6, 5) | 0.06 (0.547) | -0.24 (0.288) | -0.41 (0.212) | -0.42 (0.440) | -0.40 (0.430)
  Day 50 (n =6, 5, 7, 7, 6) | 0.15 (0.769) | -0.08 (0.335) | -0.24 (0.326) | -0.33 (0.754) | -0.40 (0.580)
Statistical Analysis 1: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg; Day 29: Repeated measures analysis of change is performed with change from baseline as dependent variable, treatment as a factor and baseline as covariate; Test type: Superiority or Other; p = 0.419, Mixed meal tolerance test; LS Mean Difference = -0.21, 80% CI 2-sided [-0.54 to 0.12], Standard Error of Mean 0.251
Statistical Analysis 2: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p = 0.077, Mixed meal tolerance test; LS Mean Difference = -0.41, 80% CI 2-sided [-0.71 to -0.12], Standard Error of Mean 0.224
Statistical Analysis 3: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p = 0.147, Mixed meal tolerance test; LS Mean Difference = -0.34, 80% CI 2-sided [-0.65 to -0.04], Standard Error of Mean 0.230
Statistical Analysis 4: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p = 0.086, Mixed meal tolerance test; LS Mean Difference = -0.43, 80% CI 2-sided [-0.76 to -0.11], Standard Error of Mean 0.244

28. Secondary Outcome: Change From Baseline in Fructosamine Levels at Day 8, 15 and 29: Stage 1
Time Frame: Baseline, Day 8, 15 and 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: micromole per liter (mcmol/L)
Groups:
- Stage 1: PF-04856883 24mg: Participants received PF-04856883 24 mg subcutaneous injection once on Day 1 in Stage 1.
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24mg | Stage 1: PF-04856883 36 mg
Number analyzed (Participants) | 15 | 5 | 6 | 6 | 7 | 5 | 7
micromole per liter (mcmol/L)
  Baseline (n =15, 5, 6, 6, 7, 5, 7) | 270.60 (34.618) | 289.20 (48.329) | 279.67 (30.507) | 304.83 (45.155) | 263.43 (34.942) | 259.80 (53.644) | 273.71 (36.036)
  Change at Day 8 (n =15, 5, 5, 6, 7, 5, 7) | 1.13 (14.461) | 20.20 (10.986) | 4.20 (18.295) | 5.67 (13.095) | 4.29 (16.720) | -13.60 (23.554) | -12.29 (10.579)
  Change at Day 15 (n =15, 5, 5, 6, 6, 5, 7) | -5.67 (17.839) | -20.40 (25.393) | -16.40 (13.502) | -9.17 (25.135) | 13.33 (24.188) | -9.60 (22.267) | -3.00 (11.165)
  Change at Day 29 (n =15, 5, 5, 6, 7, 5, 7) | 0.93 (19.627) | 8.40 (30.876) | 7.20 (29.660) | -4.50 (16.109) | 15.86 (24.024) | 1.40 (17.344) | -4.43 (18.867)

29. Secondary Outcome: Change From Baseline in Fructosamine Levels at Day 8, 15, 22, 29 and 50: Stage 2
Time Frame: Baseline, Day 8, 15, 22, 29 and 50
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 7 | 5 | 7 | 7 | 6
mcmol/L
  Baseline (n =7, 5, 7, 7, 6) | 281.14 (57.875) | 309.40 (47.600) | 301.14 (43.690) | 291.29 (37.911) | 303.67 (47.272)
  Change at Day 8 (n =7, 5, 7, 6, 6) | -5.29 (19.678) | -8.20 (11.100) | -12.14 (12.668) | -9.17 (23.043) | -10.17 (21.720)
  Change at Day 15 (n =7, 5, 7, 6, 6) | -1.86 (21.146) | -8.20 (15.707) | -39.29 (21.077) | -11.67 (24.047) | -14.67 (33.037)
  Change at Day 22 (n =7, 5, 7, 6, 6) | -7.43 (13.176) | -18.20 (20.462) | -37.86 (19.945) | -24.67 (20.925) | -27.50 (25.399)
  Change at Day 29 (n =7, 5, 7, 6, 4) | -4.43 (27.098) | -26.60 (22.612) | -37.57 (14.976) | -32.67 (28.507) | -41.00 (29.855)
  Change at Day 50 (n =7, 5, 7, 7, 6) | -6.86 (20.732) | -8.80 (14.446) | -6.43 (20.871) | -12.43 (26.732) | -5.67 (31.258)
Statistical Analysis 1: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg; Day 8: Repeated measures analysis of change is performed with change from baseline as dependent variable, treatment as a factor and baseline as covariate; Test type: Superiority or Other; p = 0.663, Mixed meal tolerance test; LS Mean Difference = 4.11, 80% CI 2-sided [-8.16 to 16.37], Standard Error of Mean 9.326
Statistical Analysis 2: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg; [analysis description as in outcome 29, analysis 1]; Test type: Superiority or Other; p = 0.825, mixed meal tolerance test; LS Mean Difference = -1.89, 80% CI 2-sided [-13.03 to 9.25], Standard Error of Mean 8.472
Statistical Analysis 3: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg; [analysis description as in outcome 29, analysis 1]; Test type: Superiority or Other; p = 0.878, Mixed meal tolerance test; LS Mean Difference = 1.36, 80% CI 2-sided [-10.20 to 12.92], Standard Error of Mean 8.791
Statistical Analysis 4: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg; [analysis description as in outcome 29, analysis 1]; Test type: Superiority or Other; p = 0.936, Mixed meal tolerance test; LS Mean Difference = 0.72, 80% CI 2-sided [-10.89 to 12.33], Standard Error of Mean 8.829
Statistical Analysis 5: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg; Day 15: Repeated measures analysis of change is performed with change from baseline as dependent variable, treatment as a factor and baseline as covariate; Test type: Superiority or Other; p = 0.959, Mixed meal tolerance test; LS Mean Difference = 0.68, 80% CI 2-sided [-16.46 to 17.82], Standard Error of Mean 13.037
Statistical Analysis 6: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg; [analysis description as in outcome 29, analysis 5]; Test type: Superiority or Other; p = 0.011, Mixed meal tolerance test; LS Mean Difference = -32.46, 80% CI 2-sided [-48.07 to -16.85], Standard Error of Mean 11.872
Statistical Analysis 7: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg; [analysis description as in outcome 29, analysis 5]; Test type: Superiority or Other; p = 0.833, Mixed meal tolerance test; LS Mean Difference = -2.61, 80% CI 2-sided [-18.67 to 13.45], Standard Error of Mean 12.212
Statistical Analysis 8: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg; [analysis description as in outcome 29, analysis 5]; Test type: Superiority or Other; p = 0.565, Mixed meal tolerance test; LS Mean Difference = -7.21, 80% CI 2-sided [-23.47 to 9.05], Standard Error of Mean 12.365
Statistical Analysis 9: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg; Day 22: Repeated measures analysis of change is performed with change from baseline as dependent variable, treatment as a factor and baseline as covariate; Test type: Superiority or Other; p = 0.703, Mixed meal tolerance test; LS Mean Difference = -3.75, 80% CI 2-sided [-16.52 to 9.02], Standard Error of Mean 9.713
Statistical Analysis 10: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg; [analysis description as in outcome 29, analysis 9]; Test type: Superiority or Other; p = 0.008, Mixed meal tolerance test; LS Mean Difference = -25.46, 80% CI 2-sided [-37.07 to -13.85], Standard Error of Mean 8.827
Statistical Analysis 11: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg; [analysis description as in outcome 29, analysis 9]; Test type: Superiority or Other; p = 0.253, Mixed meal tolerance test; LS Mean Difference = -10.60, 80% CI 2-sided [-22.51 to 1.32], Standard Error of Mean 9.061
Statistical Analysis 12: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg; [analysis description as in outcome 29, analysis 9]; Test type: Superiority or Other; p = 0.128, Mixed meal tolerance test; LS Mean Difference = -14.47, 80% CI 2-sided [-26.57 to -2.38], Standard Error of Mean 9.198
Statistical Analysis 13: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p = 0.196, Mixed meal tolerance test; LS Mean Difference = -15.15, 80% CI 2-sided [-30.17 to -0.13], Standard Error of Mean 11.421
Statistical Analysis 14: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p = 0.012, Mixed meal tolerance test; LS Mean Difference = -28.17, 80% CI 2-sided [-41.84 to -14.51], Standard Error of Mean 10.393
Statistical Analysis 15: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p = 0.047, Mixed meal tolerance test; LS Mean Difference = -22.48, 80% CI 2-sided [-36.65 to -8.32], Standard Error of Mean 10.773
Statistical Analysis 16: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p = 0.023, Mixed meal tolerance test; LS Mean Difference = -28.63, 80% CI 2-sided [-44.19 to -13.06], Standard Error of Mean 11.837
Statistical Analysis 17: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg; Day 50: Repeated measures analysis of change is performed with change from baseline as dependent variable, treatment as a factor and baseline as covariate; Test type: Superiority or Other; p = 0.711, Mixed meal tolerance test; LS Mean Difference = 5.08, 80% CI 2-sided [-12.77 to 22.93], Standard Error of Mean 13.576
Statistical Analysis 18: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg; [analysis description as in outcome 29, analysis 17]; Test type: Superiority or Other; p = 0.666, Mixed meal tolerance test; LS Mean Difference = 5.40, 80% CI 2-sided [-10.86 to 21.66], Standard Error of Mean 12.365
Statistical Analysis 19: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg; [analysis description as in outcome 29, analysis 17]; Test type: Superiority or Other; p = 0.807, Mixed meal tolerance test; LS Mean Difference = -3.05, 80% CI 2-sided [-19.27 to 13.17], Standard Error of Mean 12.333
Statistical Analysis 20: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg; [analysis description as in outcome 29, analysis 17]; Test type: Superiority or Other; p = 0.603, Mixed meal tolerance test; LS Mean Difference = 6.79, 80% CI 2-sided [-10.15 to 23.72], Standard Error of Mean 12.877

30. Secondary Outcome: Change From Baseline in 1, 5 Anhydroglucitol at Day 8, 15 and 29: Stage 1
Time Frame: Baseline, Day 8, 15 and 29
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg
Number analyzed (Participants) | 15 | 5 | 6 | 6 | 7 | 5 | 7
microgram per milliliter (mcg/mL)
  Baseline (n =15, 5, 6, 6, 7, 5, 7) | 8.17 (5.021) | 5.02 (2.831) | 5.77 (1.306) | 5.35 (3.683) | 6.20 (5.440) | 12.04 (5.133) | 11.84 (8.122)
  Change at Day 8 (n =15, 5, 5, 6, 7, 5, 7) | 0.39 (0.895) | -0.36 (0.727) | 0.64 (0.639) | 0.15 (0.596) | 0.73 (0.632) | 0.00 (1.584) | 0.97 (0.629)
  Change at Day 15 (n =15, 5, 5, 6, 6, 5, 7) | 0.38 (1.047) | 0.42 (1.711) | 1.50 (1.321) | -0.32 (1.143) | 1.07 (1.111) | 0.32 (1.608) | 1.17 (0.780)
  Change at Day 29 (n =15, 5, 5, 6, 7, 5, 7) | 0.46 (1.608) | -0.36 (0.820) | -0.52 (3.192) | -0.62 (1.492) | 0.97 (1.467) | 0.36 (1.499) | 0.66 (1.110)

31. Secondary Outcome: Change From Baseline in 1, 5 Anhydroglucitol at Day 8, 15, 22, 29 and 50: Stage 2
Time Frame: Baseline, Day 8, 15, 22, 29 and 50
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Stage 2: Placebo | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 7 | 5 | 7 | 7 | 6
mcg/mL
  Baseline (n =7, 5, 7, 7, 6) | 7.66 (4.351) | 6.32 (3.517) | 8.09 (6.240) | 7.59 (5.538) | 3.95 (1.291)
  Change at Day 8 (n =7, 5, 7, 6, 6) | -0.10 (0.663) | 0.40 (0.962) | 0.41 (0.570) | -0.08 (1.599) | 0.90 (0.502)
  Change at Day 15 (n =7, 5, 7, 6, 6) | -0.03 (1.376) | 0.72 (1.512) | 1.21 (0.641) | 0.32 (2.483) | 0.63 (1.481)
  Change at Day 22 (n =7, 5, 7, 6, 6) | 0.13 (1.289) | 1.14 (0.518) | 1.73 (1.034) | 0.95 (3.086) | 1.28 (2.046)
  Change at Day 29 (n =7, 5, 7, 6, 5) | 0.36 (1.765) | 1.46 (0.730) | 1.83 (1.241) | 1.50 (2.900) | 1.60 (2.827)
  Change at Day 50 (n =7, 5, 7, 7, 6) | 0.40 (2.106) | 0.38 (2.381) | -0.30 (1.294) | 1.64 (2.985) | 0.92 (2.076)
Statistical Analysis 1: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg; [analysis description as in outcome 29, analysis 1]; Test type: Superiority or Other; p = 0.387, Mixed meal tolerance test; LS Mean Difference = 0.48, 80% CI 2-sided [-0.24 to 1.21], Standard Error of Mean 0.551
Statistical Analysis 2: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg; [analysis description as in outcome 29, analysis 1]; Test type: Superiority or Other; p = 0.309, Mixed meal tolerance test; LS Mean Difference = 0.52, 80% CI 2-sided [-0.14 to 1.18], Standard Error of Mean 0.501
Statistical Analysis 3: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg; [analysis description as in outcome 29, analysis 1]; Test type: Superiority or Other; p = 0.956, Mixed meal tolerance test; LS Mean Difference = -0.03, 80% CI 2-sided [-0.71 to 0.65], Standard Error of Mean 0.518
Statistical Analysis 4: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg; [analysis description as in outcome 29, analysis 1]; Test type: Superiority or Other; p = 0.089, Mixed meal tolerance test; LS Mean Difference = 0.96, 80% CI 2-sided [0.24 to 1.67], Standard Error of Mean 0.542
Statistical Analysis 5: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg; [analysis description as in outcome 29, analysis 5]; Test type: Superiority or Other; p = 0.434, Mixed meal tolerance test; LS Mean Difference = 0.73, 80% CI 2-sided [-0.48 to 1.95], Standard Error of Mean 0.923
Statistical Analysis 6: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg; [analysis description as in outcome 29, analysis 5]; Test type: Superiority or Other; p = 0.150, Mixed meal tolerance test; LS Mean Difference = 1.25, 80% CI 2-sided [0.14 to 2.35], Standard Error of Mean 0.841
Statistical Analysis 7: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg; [analysis description as in outcome 29, analysis 5]; Test type: Superiority or Other; p = 0.752, Mixed meal tolerance test; LS Mean Difference = 0.27, 80% CI 2-sided [-0.86 to 1.41], Standard Error of Mean 0.861
Statistical Analysis 8: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg; [analysis description as in outcome 29, analysis 5]; Test type: Superiority or Other; p = 0.492, Mixed meal tolerance test; LS Mean Difference = 0.62, 80% CI 2-sided [-0.55 to 1.79], Standard Error of Mean 0.888
Statistical Analysis 9: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg; [analysis description as in outcome 29, analysis 9]; Test type: Superiority or Other; p = 0.358, Mixed meal tolerance test; LS Mean Difference = 1.00, 80% CI 2-sided [-0.40 to 2.40], Standard Error of Mean 1.064
Statistical Analysis 10: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg; [analysis description as in outcome 29, analysis 9]; Test type: Superiority or Other; p = 0.110, Mixed meal tolerance test; LS mean Difference = 1.60, 80% CI 2-sided [0.33 to 2.88], Standard Error of Mean 0.970
Statistical Analysis 11: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg; [analysis description as in outcome 29, analysis 9]; Test type: Superiority or Other; p = 0.461, Mixed meal tolerance test; LS mean Difference = 0.74, 80% CI 2-sided [-0.56 to 2.05], Standard Error of Mean 0.993
Statistical Analysis 12: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg; [analysis description as in outcome 29, analysis 9]; Test type: Superiority or Other; p = 0.286, Mixed meal tolerance test; LS mean Difference = 1.11, 80% CI 2-sided [-0.23 to 2.45], Standard Error of Mean 1.021
Statistical Analysis 13: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p = 0.362, Mixed meal tolerance test; LS Mean Difference = 1.09, 80% CI 2-sided [-0.45 to 2.63], Standard Error of Mean 1.172
Statistical Analysis 14: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p = 0.179, Mixed meal tolerance test; LS Mean Difference = 1.48, 80% CI 2-sided [0.07 to 2.88], Standard Error of Mean 1.069
Statistical Analysis 15: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p = 0.342, Mixed meal tolerance test; LS Mean Difference = 1.06, 80% CI 2-sided [-0.38 to 2.49], Standard Error of Mean 1.092
Statistical Analysis 16: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p = 0.272, Mixed meal tolerance test; LS Mean Difference = 1.27, 80% CI 2-sided [-0.22 to 2.75], Standard Error of Mean 1.129
Statistical Analysis 17: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg; [analysis description as in outcome 29, analysis 17]; Test type: Superiority or Other; p = 0.979, Mixed meal tolerance test; LS Mean Difference = -0.04, 80% CI 2-sided [-1.77 to 1.70], Standard Error of Mean 1.317
Statistical Analysis 18: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg; [analysis description as in outcome 29, analysis 17]; Test type: Superiority or Other; p = 0.568, Mixed meal tolerance test; LS Mean Difference = -0.70, 80% CI 2-sided [-2.27 to 0.88], Standard Error of Mean 1.201
Statistical Analysis 19: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg; [analysis description as in outcome 29, analysis 17]; Test type: Superiority or Other; p = 0.311, Mixed meal tolerance test; LS Mean Difference = 1.24, 80% CI 2-sided [-0.34 to 2.82], Standard Error of Mean 1.201
Statistical Analysis 20: Comparison: Stage 2: Placebo vs Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg; [analysis description as in outcome 29, analysis 17]; Test type: Superiority or Other; p = 0.710, Mixed meal tolerance test; LS Mean Difference = 0.47, 80% CI 2-sided [-1.18 to 2.13], Standard Error of Mean 1.260

32. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA): Stage 1
Time Frame: Day 1 and 29
Population: Safety population included all participants who received at least 1 dose of study medication. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Number; unit: participants
Arm/Group | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg
Number analyzed (Participants) | 5 | 6 | 6 | 7 | 5 | 7
participants
  Day 1 (n =5, 6, 6, 7, 5, 7) | 1 | 1 | 0 | 0 | 0 | 2
  Day 29 (n =5, 5, 6, 6, 5, 7) | 1 | 2 | 1 | 0 | 0 | 2

33. Secondary Outcome: Number of Participant With Anti-Drug Antibodies (ADA): Stage 2
Time Frame: Day 1, 29 and 50
Population: as for outcome 32
Measure: Number; unit: participants
Arm/Group | Stage 2: PF-04856883 12 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Number analyzed (Participants) | 5 | 7 | 7 | 6
participants
  Day 1 (n =5, 7, 7, 6) | 0 | 1 | 1 | 0
  Day 29 (n =5, 7, 6, 5) | 0 | 2 | 2 | 1
  Day 50 (n =5, 7, 6, 6) | 0 | 3 | 2 | 3

ADVERSE EVENTS:
Groups:
- Stage 2: PF-04856883 12.0 mg: Participants received single dose of PF-04856883 12.0 mg subcutaneous injection on Day 1, 8, 15 and 22 in Stage 2.
Arm/Group | Stage 1: PF-04856883 Placebo | Stage 1: PF-04856883 4 mg | Stage 1: PF-04856883 8 mg | Stage 1: PF-04856883 12 mg | Stage 1: PF-04856883 18 mg | Stage 1: PF-04856883 24 mg | Stage 1: PF-04856883 36 mg | Stage 2: Placebo | Stage 2: PF-04856883 12.0 mg | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/5 | 0/6 | 0/6 | 0/7 | 0/5 | 0/7 | 0/7 | 0/5 | 0/7 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 8/15 | 1/5 | 0/6 | 2/6 | 4/7 | 3/5 | 4/7 | 4/7 | 5/5 | 5/7 | 5/7 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: PF-04856883 Placebo (N=15) | Stage 1: PF-04856883 4 mg (N=5) | Stage 1: PF-04856883 8 mg (N=6) | Stage 1: PF-04856883 12 mg (N=6) | Stage 1: PF-04856883 18 mg (N=7) | Stage 1: PF-04856883 24 mg (N=5) | Stage 1: PF-04856883 36 mg (N=7) | Stage 2: Placebo (N=7) | Stage 2: PF-04856883 12.0 mg (N=5) | Stage 2: PF-04856883 12 mg + 12 mg + 24 mg + 24 mg (N=7) | Stage 2: PF-04856883 8 mg + 8 mg + 16 mg + 24 mg (N=7) | Stage 2: PF-04856883 12 mg + 20 mg + 28 mg + 36 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 2 | 3
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 3 | 2 | 2 | 3 | 2 | 3 | 4 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 2 | 2 | 2 | 3 | 3
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 4 | 3 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Faecal volume increased (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.